CLINICAL TRIAL: NCT04171271
Title: Effects of Motor Imagery on Autonomic Function and Motor Imagery Abilities in Healthy Individuals
Brief Title: Effects of Motor Imagery on Autonomic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-GOKAE-1150
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Motor Imagery Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Activating kinesthetic motor imagery training (Experimental)
  Interventions: Behavioral: Activating kinesthetic motor imagery training
- Relaxing kinesthetic motor imagery training (Active Comparator)
  Interventions: Behavioral: Relaxing kinesthetic motor imagery training
- Control (no specific intervention) (No Intervention)

INTERVENTIONS:
Behavioral: Activating kinesthetic motor imagery training — Participants in the activating kinesthetic motor imagery training group will imagine high effort exercises (e.g. planking, boxing, jumping, squats, push-ups) in the sessions in home using the study audio-video motor imagery script for 5 times per week; 17 min per day for 2 weeks. Phone calls will be performed for support and as a reminder for the assessment (after one week).
  Arms: Activating kinesthetic motor imagery training
Behavioral: Relaxing kinesthetic motor imagery training — Participants in the relaxing kinesthetic motor imagery training group will imagine relaxing (low effort) exercises (e.g. breathing exercises, stretching, body awareness exercises) in home using the study audio-video motor imagery script 5 times per week; 17 min per day for 2 weeks. Phone calls will be performed for support and as a reminder for the assessment (after one week).
  Arms: Relaxing kinesthetic motor imagery training

SUMMARY:
Most studies on motor imagery suggested the effects of motor imagery are related to neuroplastic changes in the brain. In addition to that the neuroplastic changes, it is thought that motor imagery can alter metabolic responses just like in actual exercise. However, the level of evidence about the effect of motor imagery on autonomic functions is limited.

The aims of this study;

1. The primary aim of this study is to investigate the effects of activating and relaxing kinesthetic motor imagery on autonomic function in healthy individuals and to compare these two methods.
2. The secondary aim of this study is to explore the effects of these methods on motor imagery skills of individuals will also be investigated.

The participants will randomly be allocated into three groups: (1) Activating kinesthetic motor imagery training, (2) Relaxing kinesthetic motor imagery training, and (3) Control group.

Participants in the activating kinesthetic motor imagery training group will imagine high effort exercises (e.g. planking, boxing, jumping, squats, push-ups) in the sessions in home using the study audio-video motor imagery script. The relaxing kinesthetic motor imagery training group will imagine relaxing (low effort) exercises (e.g. breathing exercises, stretching, body awareness exercises) in home using the study audio-video motor imagery script. Prior the sessions, the participants will receive an introductory lecture about motor imagery. The intervention groups will practise 5 times per week for 17 minutes per day for 2 weeks. Phone calls will be performed for support and as a reminder for the assessment (after one week). The control group will receive no specific training. Data will be collected at baseline and after the two-week intervention by masked outcome assessors.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy (not having any known chronic disease)
* Volunteer to participate in the study

Exclusion Criteria:

* Pregnancy
* Previous disorder/surgery history that can alter physical performance

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the methods - minimum recruitment rate | through Study Completion, an Average of 8 Months
  A minimum recruitment rate of 10 participants per month will be accepted as feasiable.
Feasibility of the methods - minimum retention rate | through Study Completion, an Average of 8 Months
  A target retention rate of 80% will be accepted as feasiable.
Feasibility of the methods - minimum adherence rate | through Study Completion, an Average of 8 Months
  A target minimum adherence rate of 70% of the overall practice sessions will be accepted as feasiable.
Feasibility of the methods - adverse events | through Study Completion, an Average of 8 Months
  A record sheet was prepared for possible adverse events during the tests and intervention. It includes information about seriousness, expectedness, severity, causality, time, duration of the event and clinical action taken. The numbers of adverse events will be reported.

SECONDARY OUTCOMES:
Edinburgh Handedness Inventory | at Baseline
  The Edinburgh Handedness Inventory is a measurement scale used to assess the dominance of a person's right or left hand in everyday activities, sometimes referred to as laterality. The 10-item inventory contains a list of instructions to be carried out by the individual being assessed. Items are rated by direct observation of the individual's behavior or by self-report of everyday behavior. Scoring is as follows: "-50" always left, "-25" usually left, "0" no preference, "25" usually right, and "50" always right. Scores on the eight rows are summed to provide a score of -400 to +400. Positive scores indicate right-hand dominance and negative scores indicate left-hand dominance.
Movement Imagery Questionnaire-Revised | Change from Baseline at 2 Weeks
  The Movement Imagery Questionnaire-Revised assesses visual and kinesthetic movement imagery ability and is comprised of four visual and four kinesthetic items. Each item entails performing a movement, visually or kinesthetically imaging that movement and then rating the ease or difficulty of generating that image on a 7-point scale from 1 = very hard to see/feel to 7 = very easy to see/feel. Higher scores indicate higher visual or kinesthetic movement imagery ability.
Mental chronometry for walking task | Change from Baseline at 2 Weeks
  The participants will actually execute and imagine a motor task: walking at comfortable speed for a distance of 6 m. The duration of actual and imagined movements will be recorded by means of an electronic stopwatch. During the execution of the actual and imagined movements subjects will hold the electronic stopwatch in their non-dominant hand. They will start the stopwatch when they started to move (actual or imagined movement) and they will stop it when they completed their movement (actual or imagined). Delta time will be calculated with the formula [(actual - imagined) / (actual + imagined / 2)] × 100. Lower scores indicate higher motor imagery ability.
Mental chronometry for writing task | Change from Baseline at 2 Weeks
  The participants will actually execute and imagine a motor task: writing the following sentence: "Türkiye'nin başkenti Ankara". The duration of actual and imagined movements will be recorded by means of an electronic stopwatch. During the execution of the actual and imagined movements subjects will hold the electronic stopwatch in their non-dominant hand. They will start the stopwatch when they started to move (actual or imagined movement) and they will stop it when they completed their movement (actual or imagined). Delta time will be calculated with the formula [(actual - imagined) / (actual + imagined / 2)] × 100. Lower scores indicate higher motor imagery ability.
Hand Laterality Judgement Measurement | Change from Baseline at 2 Weeks
  A tablet including an application Recognise™ app, NOI) will be placed on a table while the participants sitting in a standard chair. When given the cue to begin, participants will view the image and touch the screen to select the appropriate hand laterality judgement image interpretation. A standard 5-s maximum time limit per image will be set on the app. At the completion of the 40 images the accuracy for right, left, and total will be recorded along with average time per image to the nearest hundredth of a second.
Resting Metabolic Rate Measurements - Oxygen Consumption | Change from Baseline at 2 Weeks
  Quark cardiopulmonary exercise testing system will be used to assess Resting Metabolic Rate Measurements. Oxygen consumption is an indicator of aerobic capacity. Higher scores indicate higher aerobic capacity.
Resting Metabolic Rate Measurements - Respiratory Exchange Ratio | Change from Baseline at 2 Weeks
  Quark cardiopulmonary exercise testing system will be used to assess Resting Metabolic Rate Measurements. The ratio of carbon dioxide output/oxygen uptake is called the respiratory exchange ratio. Under steady state conditions, the respiratory exchange ratio equals the respiratory quotient. The respiratory quotient value is determined by the fuels used for metabolic processes. An respiratory quotient of 1 indicates metabolism primarily of carbohydrates, whereas an respiratory quotient of <1 indicates a mixture of carbohydrates and fat (respiratory quotient about 0.7) or protein (respiratory quotient about 0.8).

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided